CLINICAL TRIAL: NCT04786704
Title: Detection of Advanced Colorectal Neoplasia for Stool DNA in Asymptomatic Chinese Population : A Multi-central Community-based Screening Study
Brief Title: A Stool DNA Test for Detection of Advanced Colorectal Neoplasia in Asymptomatic Chinese Community Population
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Gongli Hospital of Shanghai Pudong New Area (Unknown); Shanghai Songjiang District Central Hospital (Unknown); Shanghai Jing'an District Central Hospital (Unknown); Tongji University (Other); Qingyuan People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); 900 Hospital of Joint Logistics Support Force of PLA (Other); First Affiliated Hospital of Suzhou Medical College (Other); Affiliated Hospital of Jiangnan University (Other); Traditional Chinese Medicine Hosipital of Kunshan (Unknown); Ankang Central Hospital (Other); Shandong Cancer Hospital and Institute (Other); Ningjin County Hospital (Unknown)
Responsible Party: Principal Investigator, Zhaoshen Li, MD,Director, Head of Department of Gastroenterology and Digestive Endoscopy Center, Principal Investigator, Clinical Professor, Changhai Hospital
Other Study IDs: SDC2_Community
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer; Colorectal Neoplasm; Advanced Adenoma; Adenoma; Serrated Lesion
Keywords: Methylated Syndecan-2(SDC2); Stool DNA; Fecal immunochemical test; Advanced colorectal neoplasia; Asia-Pacific Colorectal Screening score
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Stool-based SDC2 DNA methylation test — A diagnostic device measuring syndecan 2(SDC2) methylation status in stool DNA to detect colorectal cancer
  Other Names: COLOSAFE
Diagnostic Test: quantitative Fecal immunochemical test — A diagnostic device using immunoturbidimetric methods to measure fecal hemoglobin concentration
  Other Names: OC-Sensor

SUMMARY:
to determine screening value of stool-based SDC2 DNA methylation test for advanced colorectal neoplasia in the asymptomatic Chinese community population.

DETAILED DESCRIPTION:
In China, colorectal cancer (CRC) remains to be the leading cancer of the digestive system. According to nationwide cancer statistics using population-based cancer registry data in China, age-standardized incidence rate of CRC and age-standardized mortality rate increased significantly from 2000 to 2015. It induces a substantial financial burden in terms of healthcare utilization and quality-adjusted life years (QALY) lost. Fecal Occult Blood Tests (FOBT) and colonoscopy have been proposed as the main primary screening modalities for asymptomatic subjects by international guidelines and Asia Pacific Consensus Statements. Nevertheless, shortage and uneven distribution of colonoscopy resources combined with huge population base consisted of the current situation in China. Previous population-based CRC screening programs usually employed questionnaires and/or FOBT to assess high-risk groups and recommended colonoscopy. This algorithm faced difficulties such as complex traditional questionnaires, low colonoscopy adherence, and a high false-positive rate. When the Coronavirus disease 2019 pandemic further limited the implementation of colonoscopy, the contradictions developed more acute.

A Hong Kong group had designed and validated a colorectal cancer risk scoring system based on age, gender, smoking history, and family history through the results of screening in 11 Asia-Pacific cities. The Asia-Pacific Colorectal Screening (APCS) score was more concise and divided the population into three categories: low risk, intermediate risk, and high risk. Compared with the low-risk population, the probability of advanced colorectal neoplasia in intermediate-risk and high-risk population increased by 2.6 times and 4.3 times respectively. Because of simplicity and efficiency, it was recommended by Asia-Pacific screening guidelines and several guidelines in China. Another APCS related multi-center study indicated that by selecting high-risk subjects and low/average-risk subjects with a positive fecal immunochemical test (FIT) for colonoscopy, the colonoscopy workload could be reduced by 50% compared with the strategy of primary colonoscopy in those same subjects. All these experiences deserved to be drawn on during the post-pandemic era.

The recent decade has witnessed a rapid development of non-invasive biomarkers to detect CRC. Stool DNA(sDNA) Testing is a novel screening test for CRC, using molecular techniques to identify CRC-relevant biomarkers in stool. One of its toolkits, Multitarget Stool DNA Testing (FIT-DNA), was first approved by the FDA in 2014 for its application in clinical practice, which has been widely promoted in the United States. Subsequently, it was endorsed by multiple societies as one of the recommended screening tests.

Recently, a stool test of methylated Syndecan-2(SDC2) has been developed as a fecal-DNA product targeted to improve the diagnostic accuracy of CRC screening. A meta-analysis of previous clinical studies reporting the accuracy of stool DNA methylation tests in detecting CRC included 46 studies totaling 16,149 patients. The most accurate single gene was found to be SDC2 with a pooled sensitivity of 83.1% (72.6%, 90.2%) and a specificity of 91.2% (88.6%, 93.2%). A recent study involving 1,110 subjects from 2017 to 2018 by three Chinese tertiary hospitals assessed the performance of the SDC2 sDNA test. The sensitivity of the SDC2 sDNA test was 301/359 (83.8%) for CRC, 16/38 (42.1%) for advanced adenomas, and 134/154 (87.0%) for early-stage CRC (stage I-II), while maintaining a specificity of 699/713 (98.0%). Nevertheless, there were limitations in the design of these original studies. For instance, most involved small, hospital-based CRC cases and controls that might not fill the knowledge gap between population screening. Additional clinical trials are required to further validate its diagnostic accuracy in other populations, especially community-setting.

Potential participates would be recruited via community public communication. The subjects would be asked to fill in a concise questionnaire obtained through a public WeChat account after informed consent. Basic information would be acquired while APCS score and correspondent risk categories would be calculated automatically. After sampling education, stool collection devices of sDNA and quantitative fecal immunochemical test (qFIT) would be distributed to all subjects. Two samples of stool from single defecation would be requested to put into the two collection devices according to instructions respectively by the subjects themselves at home.

Efforts would be made by the public WeChat account and the community staff to urge samples recover from subjects as quickly as possible (prefer within 24h after defecation). Community staff would deliver the samples qualified in the initial evaluation to the standardized laboratory for testing as quickly as possible. If APCS be evaluated high-risk or any of qFIT or sDNA tests positive, the risk of the subject would be considered increased. Colonoscopy would be strongly recommended, and priority and rapid arrangement would be made in the corresponding center. For subjects with low/intermediate-risk APCS and negative qFIT and sDNA, the project team also encourages the subjects to accept colonoscopy on the basis of a clear understanding of benefits and risks. We would help to arrange colonoscopy as early as possible.

All colonoscopy examinations will be performed by experienced endoscopists while monitoring quality of colonoscopy (bowel preparation, cecal intubation rate and withdrawal time). Full-time recording personnel would be arranged to follow up and record the relevant information of colonoscopy. For the subjects diagnosed with colorectal cancer, the postoperative diagnosis and tumor-node-metastasis (TNM) staging of the subjects would be retrieved.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic screening individual (no alarm features predicting colorectal cancer including hematochezia, melena, anemia of unknown cause, weight loss, abdominal mass, a positive result of digital rectal examination)
2. Age between 45 to 75 years old, the gender is not limited
3. Willing to participate and sign informed consent

Exclusion Criteria:

1. Patients with contraindications for bowel preparation or colonoscopy
2. Patients with known colorectal adenoma or serrated lesions
3. History of colonoscopy within 5 years or polypectomy
4. Patients with inflammatory bowel disease
5. History of CRC and patients clinically highly suspected with colorectal cancer
6. History of hereditary CRC syndrome (including polyposis)
7. Patients taking anticoagulants such as aspirin and warfarin within 7 days, or who have coagulopathy
8. Pregnancy, or severe organ insufficiency (heart, lung, or kidney et al)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community residents were invited to participate in the evaluation. All the individuals involved would undergo APCS evaluation, qFIT, and sDNA tests. A participator would be considered with increased CRC risk if any of the three is evaluated high-risk or tested positive and would be subsequently recommended to receive timely colonoscopy. When the APCS evaluation shows low or Intermediate risk with both negative results of qFIT and sDNA, participators would be encouraged to undergo colonoscopy based on patient preferences, which could also provide a refference for the prevanlence of advanced colorectal neoplasia in low-risk patients.
Sampling Method: Non-Probability Sample
Enrollment: 12106 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Detection of advanced colorectal neoplasia | Through study completion, an average of 1 year
  Advanced colorectal neoplasia is defined as a colorectal adenoma or sessile serrated lesion ≥10 mm, adenoma or sessile serrated lesion with tubulovillous or villous histology, adenoma with high-grade dysplasia, traditional serrated adenoma, or presence of colorectal cancer.

SECONDARY OUTCOMES:
Compliance rate of colonoscopy | Through study completion, an average of 1 year
  The compliance rate of colonoscopy was calculated as the number of recieving colonoscopy divdied the number of accomplishing primary evaluation of APCS, stool DNA or FIT.
Detection of colorectal cancer | Through study completion, an average of 1 year
  Lesions will be confirmed as malignant by histopathologic examination.
Detection of colorectal neoplasia | Through study completion, an average of 1 year
  Advanced colorectal neoplasia is defined as a colorectal adenoma or sessile serrated lesion, traditional serrated adenoma, hyperplastic polyp ≥10 mm, or colorectal cancer.
  Lesions will be confirmed as malignant or precancerous by histopathologic examination.
Efficacy of sDNA in the detection of advanced colorectal neoplasia in high-risk asymptomatic subgroup. | Through study completion, an average of 1 year
  High-risk subgroup: APCS calculated high-risk or qFIT positive. A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination.
Efficacy of sDNA in the detection of advanced colorectal neoplasia in low-risk asymptomatic subgroup. | Through study completion, an average of 1 year
  Low-risk subgroup: APCS calculated low or medium risk, and qFIT negative. A diagnostic colonoscopy procedure is the reference method. Lesions will be confirmed as malignant or precancerous by histopathologic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, MD, Principal Investigator — Changhai Hospital, Navy/Second Military Medical University
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niu F, Wen J, Fu X, Li C, Zhao R, Wu S, Yu H, Liu X, Zhao X, Liu S, Wang X, Wang J, Zou H. Stool DNA Test of Methylated Syndecan-2 for the Early Detection of Colorectal Neoplasia. Cancer Epidemiol Biomarkers Prev. 2017 Sep;26(9):1411-1419. doi: 10.1158/1055-9965.EPI-17-0153. Epub 2017 Jun 15. PMID 28619831
- [Background] Wang J, Liu S, Wang H, Zheng L, Zhou C, Li G, Huang R, Wang H, Li C, Fan X, Fu X, Wang X, Guo H, Guan J, Sun Y, Song X, Li Z, Mu D, Sun J, Liu X, Qi Y, Niu F, Chen C, Wu X, Wang X, Song X, Zou H. Robust performance of a novel stool DNA test of methylated SDC2 for colorectal cancer detection: a multicenter clinical study. Clin Epigenetics. 2020 Oct 30;12(1):162. doi: 10.1186/s13148-020-00954-x. PMID 33126908
- [Background] Gachabayov M, Lebovics E, Rojas A, Felsenreich DM, Latifi R, Bergamaschi R. Performance evaluation of stool DNA methylation tests in colorectal cancer screening: a systematic review and meta-analysis. Colorectal Dis. 2021 May;23(5):1030-1042. doi: 10.1111/codi.15521. Epub 2021 Jan 25. PMID 33410272
- [Background] Yeoh KG, Ho KY, Chiu HM, Zhu F, Ching JY, Wu DC, Matsuda T, Byeon JS, Lee SK, Goh KL, Sollano J, Rerknimitr R, Leong R, Tsoi K, Lin JT, Sung JJ; Asia-Pacific Working Group on Colorectal Cancer. The Asia-Pacific Colorectal Screening score: a validated tool that stratifies risk for colorectal advanced neoplasia in asymptomatic Asian subjects. Gut. 2011 Sep;60(9):1236-41. doi: 10.1136/gut.2010.221168. Epub 2011 Mar 14. PMID 21402615
- [Background] Chiu HM, Ching JY, Wu KC, Rerknimitr R, Li J, Wu DC, Goh KL, Matsuda T, Kim HS, Leong R, Yeoh KG, Chong VH, Sollano JD, Ahmed F, Menon J, Sung JJ; Asia-Pacific Working Group on Colorectal Cancer. A Risk-Scoring System Combined With a Fecal Immunochemical Test Is Effective in Screening High-Risk Subjects for Early Colonoscopy to Detect Advanced Colorectal Neoplasms. Gastroenterology. 2016 Mar;150(3):617-625.e3. doi: 10.1053/j.gastro.2015.11.042. Epub 2015 Nov 25. PMID 26627608